CLINICAL TRIAL: NCT00256074
Title: The Effects of Nutritional Support of Critically Ill Patients Requiring Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision was made to terminate the project due to slower than anticipated recruitment and many of the investigators no longer being available.
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.263
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy Group (Other): Standard therapy group. Will receive high carbohydrate, low fat enteral feeding, (16.7% protein, 30% fat and 53.3% carbohydrate). The target rate is determined by the treating physician and dietician, for a minimum of 5 days following randomisation.
  Interventions: Procedure: Enteral feeding formula
- Alternative Therapy Group (Other): 2.Alternative therapy group will receive high-fat, low carbohydrate enteral feeding, (16.7% protein, 55.2% fat and 28.1% carbohydrates. At a target rate determined by the treating physician and dietician, for a maximum of 5 days following randomisation.
  Interventions: Procedure: Enteral feeding formula

INTERVENTIONS:
Procedure: Enteral feeding formula

SUMMARY:
The purpose of this study is to assess the impact of different feeding solutions on patients with breathing difficulty being supported by a breathing machine.

The aim of the study is to determine if high fat-low carbohydrate feeding reduces the carbon dioxide production in patients with respiratory failure.

DETAILED DESCRIPTION:
Patients who agree to participate in the study and fulfil the inclusion criteria, will be randomised to one of two treatment groups.

1. Standard therapy group. Will receive high carbohydrate, low fat enteral feeding, (16.7% protein, 30% fat and 53.3% carbohydrate). The target rate is determined by the treating physician and dietician, for a minimum of 5 days following randomisation.
2. Alternative therapy group will receive high-fat, low carbohydrate enteral feeding, (16.7% protein, 55.2% fat and 28.1% carbohydrates. At a target rate determined by the treating physician and dietician, for a maximum of 5 days following randomisation.

All patients will receive enteral feeding by continuous flow for 24 hours a day. The decision to commence or cease enteral feeding will remain with the treating physician.

The measurement of VO2, VCO2, resting energy expenditure and respiratory quotient wil be made on all participants 12 hourly for a maximum of 5 days using the direct calorimeter. The indirect calorimeter is connected to the expiratory outlet of the ventilator, collecting and analyzing gas that is normally discharged in to the atmosphere.

The hypothesis of the study is that the use of high- fat, low-carbohydrate enteral feed, significantly reduces the carbon dioxide production and the respiratory quotient in critically ill, mechanically ventilated patients with respiratory failure. Compared to standard high-carbohydrate low-fat enteral feed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, 18 years or older admitted with acute respiratory failure (PaO2/FiO2 <300), needing mechanical ventilation. Are expected to be require mechanical ventilation for more than 48 hours.
2. Patients who are to receive enteral feeding via a gastric or post-pyloric feeding tube.
3. Patients or their next-of-kin consent to participate in the study. -

Exclusion Criteria:

1. Patients under the age of 18 years
2. Patients with contra-indications to enteral feeding
3. Patients receiving total parental nutrition
4. Patients who are already enrolled in another study that may influence the outcome of this study.
5. Patients who are not receiving active medical management or are expected to die within 24 hours at the time of study entry.
6. Patients with diabetes mellitus, renal failure or liver failure.
7. Patients or next-of-kin who do not consent to participate in the study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine if high-fat low-carbohydrate enteral feeding reduces the carbon dioxide production and the respiratory quotient in patients with respiratory failure. | patients will be followed until death or hospital discharge

SECONDARY OUTCOMES:
1. If high-fat, low-carbohydrate enteral feeding reduces carbon dioxide production, dead space ventilation the number of days spent on mechanical ventilation,or the length of ICU stay, hospital length of stay or mortality. | patients will be followed until death or hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Megan Robertson, MBBS, Principal Investigator — Melbourne Health
Locations (1):
- Intensive Care Unit, The Royal Melbourne Hospital,, Parkville, Victoria, Australia